Official Title: An Acceptance Based PrEP Intervention to Engage Young Black MSM in the

South

NCT Number: NCT05087680

**Document Date:** 09/14/2023

# **ACTPrEP Intervention**

| ACTPrEP Int |
|---------------------------------------------------------------------|
| Session Content |
| Session 1 Outline (60 minutes) |
| 1. Introduce self, review goal of study, review confidentiality [5] |
| mins] |
| 2. Primary Values Exercise [15 minutes] |
| 3. PrEP Education (Psychoeducation) [2.5 mins] |
| □ What is PrEP |
| 4. PrEP is Prevention & Similar to Other Medications |
| (Alternative Perspective Taking) [2.5 minutes] |
| 5. Carrying Weight Metaphor: Control in Reducing HIV Risk |
| (Acceptance) [5 minutes} |
| 6. Discuss Barriers to PrEP Use [10 minutes] |
| 7. Coffee Cup Experiential Exercise (Alternative Perspective |
| Taking) [5 minutes] |
| 8. 5-Year-Old Self (Self-Compassion) [5 minutes] |
| 9. Action Plan & End of Session [5 minutes] |
| Session 2 Outline (35-45 minutes) |
| 1. Review previous session [5 minutes] |
| 2. PrEP Education (Psychoeducation) & TEAMS [5 minutes] |
| □ Forms of PrEP & PrEP Safety (PrEP & HIV medications are |
| the same/long term side effects) |
| 3. Lack of Control: Emotion Machine (Acceptance) [5 minutes] |
| 4. Cost of Avoiding Emotions Related to PrEP: Select Between 2 |
| Lives (Acceptance) [5 minutes] |
| 5. Singing Thoughts: Coping with Anxious Thoughts (Defusion) |
| [5 minutes] |
| 6. Coping with Emotions Using Senses (Present Moment |
| Awareness) [5 minutes] |
| 7. Action Plan & End of Session [5 minutes] |
| Session 3 Outline (35-45 minutes) |
| 1. Review previous session [5 minutes] |
| 2. Dimensions of Sexuality (Psychoeducation, Acceptance) [10 |
| minutes] |
| 3. Influential People and Aspired Qualities (Values) [5 minutes] |
| 4. Health of Others-Putting on Your Mask First (Values) [5 |
| minutes] |
| 5. Annoying Cousin at Party: Alternative to Controlling |
| Thoughts and Emotions [5 minutes] |
| 6. Car Self-Worth Metaphor (Acceptance, Compassion, Self as |
| Context) [5 minutes] |
| 7. Honoring Past, Future, and Present Peers Exercise (Values and |
| Perspective Taking) [5 minutes] |
| 8 Fnd of Session [5 minutes] |

8.End of Session [5 minutes]

| Session | Key Message |
|---|---|
| Number | Key Wessage |
| Session<br>One | <ul> <li>Define Values &amp; Select Individual Values</li> <li>Provide Brief PrEP Psychoeducation</li> <li>New Frame of Reference/Alternative Perspective Taking (PrEP Similar to Antibiotics)</li> <li>Acceptance of HIV Risk</li> <li>Identify &amp; Address Barriers to PrEP Use</li> <li>New Frame of Reference/Alternative Perspective Taking (Control of Health)</li> <li>Self-Compassion Exercise</li> <li>Identify Values Consistent Behaviors</li> </ul> |
| Session<br>Two | <ul> <li>Problem Solve Engaging in Values Consistent Behaviors</li> <li>Discuss PrEP Side Effects &amp; Normalize Anxiety Related to Side Effects</li> <li>Identify TEAMS Related to PrEP Side Effects</li> <li>Acceptance of Unwanted TEAMS</li> <li>Discuss Cost of Trying to Control Unwanted Thoughts and Emotions</li> <li>Identify Additional Values Consistent Behaviors</li> </ul> |
| Session<br>Three | <ul> <li>Further Define Values (Related to Influential People)</li> <li>Acceptance: Cost of Controlling Unwanted Experiences &amp; Alternative Behaviors to Controlling Thoughts and Emotions</li> <li>New Frame of Reference/Alternative Perspective Taking (PrEP Use to Honor Community &amp; Past Peers)</li> <li>Identify Additional Values Consistent Behaviors</li> </ul> |

#### **Intervention Manual**

#### **Session One**

#### **Session 1 Outline (60 minutes)**

- 1.Introduce self, review goal of study, review confidentiality [5 mins]
- 2.Primary Values Exercise [15 minutes]
- 3.PrEP Education (Psychoeducation) [2.5 mins]
  - □ What is PrEP
- 4.PrEP is Prevention & Similar to Other Medications (Alternative Perspective Taking)[2.5 minutes]
- 5. Carrying Weight Metaphor: Control in Reducing HIV Risk (Acceptance) [5 minutes]
- 6.Discuss Structural Barriers to PrEP Use [10 minutes]
- 7. Coffee Cup Experiential Exercise (Alternative Perspective Taking) [5 minutes]
- 8. Hand on Heart Exercise (Self-Compassion) [5 minutes]
- 9. Action Plan & End of Session [5 minutes]

#### Introductions

- Introduce yourself and your job/role.
- Share some information about how this work is meaningful to the interventionist, perhaps a piece of personal history regarding this work or the value of this work to the interventionist.
- Thank the participant for completing the survey and participating in the study.
- Review the goal of the study.
- Remind participant that of confidentiality and its limits.

Hi, my name is \_\_\_\_\_ and I work as a \_\_\_\_ at \_\_\_\_. Thank you for completing the survey and for your willingness to participate in this study session. The goal of this study is to understand what your thoughts and attitudes are about PrEP and to explore with you how PrEP might, or might not, fit with your life. Anything you say during this meeting will be kept confidential and not shared with anyone else. The only exception to this is if you were to report thoughts and intent of harming yourself or someone else, the law requires that we speak about these things to protect you and other folks.

We will be audio recording these sessions so that our study team can be sure I covered all the topics. All recordings are saved on a secure drive and will not be linked back to your name. Basically, when we finish today, I will listen to it and I will go through and check a box, yes, we covered this, yes, we covered this, and then we will delete it. Any questions before we get started?

#### Primary Values Exercise (Values)

Our first exercise today will be discussing what is important to you. For most of us, we live our life based on routine. We may not know why we do the things we do. Values are our heart's deepest desires for the way we want to live. They motivate us as we move through life. Values are directions we keep moving in, whereas goals are what we want to achieve along the way. For example, if you want to be a loving, caring, supportive partner, that is a value – an ongoing process. You don't just get to buy your husband chocolate and then check off the list, "Oh! I am

a good husband for the rest of my life," it is something that you are continuously working towards.

We are going to discuss different life areas and explore what is important within each of these life areas to you specifically.

Directions: Go through each life area. Only provide examples if patient is unable to come up with their own responses without example.

#### **Reminder Probes for all Questions:**

What does that look like? Can you describe it for me? What does that mean to you? What would that look like behaviorally? If I were watching you in a movie, how would you want me to describe your character? Why is this important?

<u>1.Relationships.</u> The first life area is within the realm of relationships. Relationships can be with anyone (your parents, relatives, friends, and co-workers). If you think about the people in your life, how do you want to be in these relationships? How would you want these individuals to describe you as a friend? What sort of labels would you want them to throw at you?

Examples: Supportive son, Attentive friend, Caring friend

**2.Health/physical well-being.** The next life area is within the realm of health and physical wellbeing. Is there anything about being healthy that is important to you or is being healthy important to you at all? Why do you want to be physically healthy? How do you want to look after your health (sleep, diet, exercise, smoking, alcohol, etc)? Why is this important? What about being healthy is important to you?

Examples: Be confident about way body looks, Live a long life, Be strong, Physically capable of living an active lifestyle, Feel good, Confidence

<u>3.Intimate Relations.</u> The next life area is with intimate relationships. What kind of partner would you like to be in a romantic relationship? How would you like your partner, boyfriend, or husband to describe you? What personal qualities would you like to have? How would you interact with your partner if you were the 'ideal you' in this relationship? Why do you think you want those things? Why would you want your partner to describe you that way?

Examples: Loving partner, Selfless partner, Passionate relationship

<u>4.Education/Work</u>: The final life area we are going to discuss is education and work. This refers to your knowledge or what kind of student or worker you want to be. This may include taking a formal class or learning via Youtube, volunteering, being a caretaker for a family member, and other forms of learning or work. What kind of student or worker do you want to be? What strengths would you like to have at work? What skills do you want to develop? What does that look like? Can you describe it for me?

Examples: Hardworking employee, Lifelong learner, Co-worker who listens, Talented worker, Successful career

# [Review the list of identified values with the participant and make edits to their values as needed. Record these values to refer back throughout the sessions].

I am documenting each of these values that you listed because they are going to come up later when we wrap up.

#### PrEP Education (Psychoeducation)

We are sort of switching gears a little bit and going into a small discussion about PrEP.

#### **Assess Participant Experience with PrEP**

Do you know what PrEP is or have you ever considered taking PrEP? [allow time for participant to respond]

#### What is PrEP

PrEP stands for preexposure prophylaxis. PrEP prevents HIV infection from spreading if you are exposed to the virus. Any person regardless of gender or age, who wants to take control of their health can benefit from PrEP.

#### PrEP is Prevention & Similar to Other Medications

There are currently three drugs used for PrEP: Truvada, Descovy, and Cabotegravir. These medications prevent HIV from spreading in individuals at risk for HIV. Other medications work in a similar way.

- ⇒ Antibiotics prior to dental procedure. Many dentists will ask you to take antibiotics a few days before a dental procedure. This helps your body get a head start fighting off any possible infections that may occur after the procedure.
- ⇒ Antiviral for cold sores. People who get cold sores on their mouth can get antiviral medication to prevent the cold sore from growing.
- ⇒ Vaccine for COVID-19. Vaccines, like the COVID-19 vaccine, are given before someone gets COVID to decrease the amount of symptoms they get.
- ⇒ **Hangover Prevention with Hydration and Ibuprofen.** Some people hydrate and take ibuprofen before heavy drinking to prevent a hangover the next day.

Have you ever had to take medication to prevent an illness or prior to a procedure to reduce risk of getting an infection?

Does it make sense that PrEP is not the only medication we take to prevent an illness?

Just like many people need preventative medications for other illnesses, folks should consider taking PrEP if:

- You sometimes have sex without using a condom OR
- You recently had a sexually transmitted infection OR
- If your partner is living with HIV OR
- You use injection drugs recreationally

Also, some medications are recommended based on geographic location and transmission rates. So just living in a certain area may indicate that certain vaccines or medications may be more useful for you. For example, the Centers for Disease Control and Prevention recommends that individuals living in or traveling to certain areas of South Africa should get the malaria vaccine to prevent contracting malaria because there are higher rates there.

- Sometimes risk is not about the behaviors we engage in but other things like genetics and where we live which are not always things we can control.
- This is also true about PrEP if you are sexually active in an area with higher rates of HIV infection, you may want to consider taking PrEP. Mississippi is among the states with the highest rates of new HIV infections. Any questions about that? Does that make sense?

The main takeaway messages from this section are that:

- PrEP is not the only medication used to prevent illness.
- Like other illnesses, PrEP may be beneficial for certain people based on where they live.

Now that you have heard about some of the risks that may make people want to take PrEP, let's think about risk in a different way.

#### Carrying Weight Metaphor: Control in Reducing HIV Risk (Acceptance)

Imagine you were born with a 500-pound weight on your shoulders (500-pounds is a lot of weight) and another person was born with 50 pounds of weight on their shoulders and you two were in a race. The rules of the game are simple – the first one to the finish line wins. Who do you think would win? Exactly! Because they have less weight to carry. This game isn't fair and although you could technically "win" the game, the game would be much harder for you if you've had the 500-pound weight. This is very similar to individuals who are at higher risk for acquiring cancer, diabetes, HIV and other health conditions. What if I offered to take 450 pounds off your shoulders to make the game even – would you take me up on my offer? Yeah, right? Nobody wants to carry 500-pounds. PrEP and other medications are like being offered the opportunity to take "weight" off your shoulders and reduce your risk of HIV and other illnesses. PrEP provides you more control of the amount of "weight" you have to experience in order to reduce HIV risk. Does this makes sense?

**Link to Values:** In the first exercise you identified (insert values identified from above). If we think about all of these values you listed, how do you think those values align with considering to take PrEP if you thought you needed PrEP? [allow time to discuss each value]

Values/Goals Mentioned in Interviews (for interventionist to refer to if needed)

- Keep community safe.
- Eliminate HIV in the community.
- Protect their partners from HIV.
- Protect themselves from HIV.

The main takeaway message from this section is that:

• HIV is similar to other illnesses like cancer, diabetes, in that you can take a medication, PrEP, to protect your health.

### Discuss Structural Barriers to PrEP Use

Can you think of anything that would get in the way of you being able to take PrEP if you decided to get a prescription? (allow patient to respond first and **then explore each barrier below**) [document which barriers the participants anticipates].

| Barrier | PrEP Resources |
|---|---|
| Finding a Doctor to<br>Prescribe PrEP | a. Open Arms Healthcare Center<br>805 E River Pl Jackson, Mississippi 39202<br>(601) 500-7660 |
| | b. Express Personal Health Jackson Medical Mall, 350 W. Woodrow Wilson Avenue. Third Floor 601-815-5861; eph@umc.edu |
| | c. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP) |
| | Primary Care Providers. |
| | a. Dr Arenia C Mallory Community Health Center |
| | 276 Nissan Pkwy Canton, Mississippi 39046<br>(601) 859-1798 |
| | b. GA Carmichael Family Health Center |
| | 1547 Jerry Clower Blvd Yazoo City, Mississippi 39194<br>(662) 746-6532 |
| | c. GA Carmichael Family Health Center |
| | 1668 W Peace St Canton, Mississippi 39046<br>(601) 859-5213 |
| | d. Jackson-Hinds Comprehensive Health Center |
| | 514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216 (601) 362-5321 |
| | e. AIDS Healthcare Foundation |
| | 766 Lakeland Dr Jackson, Mississippi 39216<br>(601) 368-3440 |
| | f. TIN $Rx$ |
| | 2657 Lakeland Dr Jackson, Mississippi 39232<br>(601) 588-2490 |
| | g. Quinn Healthcare PLLC |
| | 768 Avery N Blvd Ridgeland, Mississippi 39157<br>(601) 487-6482 |
| | h. Southern Medical Care |
| | 6600 US Highway 98, Hattiesburg, MS 39402<br>(601)-261-2727 |

| | Local Health Department (can do labs and set you up with Telehealth appointment for PrEP) You can search for providers on this website: <a href="https://www.pleaseprepme.org">https://www.pleaseprepme.org</a> |
|---|---|
| Telehealth Services | a. Jackson-Hinds Comprehensive Health Center 514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216 (601) 362-5321 b. Dr Arenia C Mallory Community Health Center 276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798 c. Open Arms Healthcare Center 805 E River Pl Jackson, Mississippi 39202 (601) 500-7660 d. Dr Arenia C Mallory Community Health Center 276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798 e. Southern Medical Care 6600 US Highway 98, Hattiesburg, MS 39402 (601)-261-2727 |
| Transportation to<br>Clinic Appointments | <ul> <li>a. Open Arms can provide transportation to appointments as long as you call and pre-schedule with the clinic.</li> <li>b. Express Personal Health does not offer transportation.</li> </ul> |
| Paying for PrEP<br>Appointments | Express Personal Health visits and labs are free. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP- Free Services) |
| Paying for PrEP<br>Medication | a. Mississippi Family Planning Waiver can cover the cost of PrEP. b. Gilead Payment Assistant Program can also help cover the cost of PrEP: https://www.am10.gilead.com/en/purpose/medication-access |
| PrEP Mailing Services | a. Jackson-Hinds Comprehensive Health Center<br>b. GA Carmichael Family Health Center<br>c. Open Arms Healthcare Center<br>d. Dr. Arenia C. Mallory Community Health Center<br>e. CVS<br>f. Walgreens |
| Adherence Techniques | a. Set an alarm on your phone b. Put your medication next to something you use everyday (toothbrush, cologne) c. Use a colorful pill box d. Ask someone to help remind you |

Many times, there will be things that get in the way or make it harder for us to live the life we want to live. We often have some unwanted experiences along the way. However, engaging in the behaviors within your control to maintain your health is the ultimate goal. We can continue to discuss how to deal with barriers later.

#### **Coffee Cup Experiential Exercise (Expect to get HIV Alternative Perspective Taking)**

Are you willing to participate in a brief exercise? [allow patient time to respond] Hold up a coffee cup or container.

What do you think is inside this cup. [allow the patient time to respond]

What else could be in this cup? [allow patient to come up with an many different options as they can]

Is there any way for you to know what is in this cup? What if I show you what the inside of the cup looks like? Now could you tell me what it is? Would you know what is inside then? [allow time for patient to respond]

Let's say you can see that it is a light brown substance. Would you know what it is then? [allow time for patient to respond]

It could still be several different things, like coffee, hot chocolate, tea. You see, there is no way of really knowing what is inside this cup until you have fully experienced and tasted what is in the cup. Life is very similar to thinking about what is inside this coffee cup. Sometimes we think we know what our future holds, even though it is not possible to know our future entirely until we have had the chance to fully experience it; not just look it, not just smell it. You've got to fully experience it. This is like how some people assume they will get HIV someday. Or some people assume they will get side effects from PrEP. Do you think it is better to assume that something awful is in this cup OR to consider all options until you have tried what is inside the cup? [allow time for patient to respond]

Remembering that there are several options available for your future, and being present to the experiences you have now, can help you decide what direction you want your life to go in and what you want to put in your life coffee cup. For example, taking a medication like PrEP to prevent HIV, not assuming that PrEP is going to cause side effects, not assuming that you are going to get HIV, or diabetes or all these other medical conditions. There are things that we can do within our control to help alleviate that. Now, the time has come to tell you what is in this cup but you'll know because you will never get to taste it.

#### The main takeaway message from this section is that:

• We shouldn't assume what the future will be. It is often unhelpful. Instead, we should do our best to take care of our health one day at a time.

#### **Child Self – Feeling Compassion (Self Compassion)**

[adapted from podcase with JoAnne Dahl, PhD]

We are going to do one last exercise before we wrap up for the day.

Slowly close your eyes and get comfortable in your seat. Begin by taking a few deep breaths. Notice how it feels to breath in and out. Notice the rise of your chest with each time you breath in and the fall as you breath out. Now, keeping your eyes closed, I want you to begin to imagine

yourself as a young child. Notice what you would be wearing as a child. What haircut you had as a child. Picture it in your mind's eye. Notice how tall you were. How many teeth you may have been missing. Just take a minute to see your child self.

Keeping your eyes closed I want you to think about what might your child self be feeling. Happiness, Sadness, Anxiety, multiple emotions. Were you carefree. Just take a second to imagine what your child self would be feeling.

Keeping your eyes closed, I want you to picture yourself today standing next to the child version of yourself. Notice how different you look now compared to then. Notice how much taller you are now. Notice how many more experiences you have now. Next, I want you to imagine what advice would you give your child self? Imagine yourself leaning down and saying this advice to your child self. After you give your child self this advice, I want you to imagine the older version of yourself giving a big hug and embracing the child version of yourself. Notice how hugging your child self makes you feel.

Take a couple more deep breathes. Slowly let the visual of your child self and older self fade away. Begin to imagine what the room looks like around you. When you are ready, no rush, you can open your eyes.

How was the exercise? What did you feel? Did you feel anything? (allow patient time to respond) The important thing to remember is that the child version of you is still in you and a part of who you are today. Just like children deserved to be loved and nurtured so does the you today deserve those things. Remember to be kind to yourself throughout each day as if you were talking to your child self. You wouldn't yell at your child self, you wouldn't guilt trip your child self (at least most folks wouldn't). You would be nice and nurture your child self.

#### **Action Plan**

We are wrapping up our session for today. Before we end, can you think of 3 action steps you can take before our next session that are in line with your values (list their values here)? [Because we are going to meet in one week, think of one thing that you can do]. It can be anything like telling your partner that you love them every day, exercising once a week, or scheduling a PrEP appointment. Something that you are not already doing that you want to build in

| scheduling a PrEP appointment. Something that you are not already doing that you want to build<br>in. |
|---|
| I |
| 2 |
| 3 |
| End of Session |
| Thank you for engaging in today's session. I would like you to review the values you identified |

Thank you for engaging in today's session. I would like you to review the values you identified once a week until we meet again. [Provide participant with their list of values and action items.] Your next appointment will be

Note: Please record values, barriers, and action items for each participant. We will use them in next session.

#### **Session Two**

#### Session 2 Outline (35 minutes)

- 1.Review previous session [5 minutes]
- 2.PrEP Education (Psychoeducation) & TEAMS [5 mins]
  - □ Forms of PrEP & PrEP Safety (PrEP & HIV medications are the same and we know long term side effects)
- 3.Lack of Control: Emotion Machine (Acceptance) [5 minutes]
- 4.Cost of Avoiding Emotions Related to PrEP: Select Between 2 Lives (Acceptance) [5 minutes]
- 5. Singing Thoughts: Coping with Anxious Thoughts (Defusion) [5 minutes]
- 6.Coping with Emotions Using Senses (Present Moment Awareness) [5 minutes]
- 5. Action Plan & End of Session [5 minutes]

#### **Review Previous Session**

Welcome back! To get started, I just want to briefly review a few things from our last session. You identified (say their values) as your values in our last session. Does that still seem accurate now that you have had time to think about things? Is there anything you would change?

You selected 3 action plan items to do that are in line with your values. How did that go? [Help participant problem solve if they were unable to complete the action plan]

How did that may you feel to complete (or not complete) the [action plan items] ?

| Action Plan |
|---|
| Similar to our last session, can you think of 3 action steps you can take before our next session that are in line with your values (list their values here)? These can be similar to the plans you listed in the last session or new ones. |
| I |
| 2. |
| 3. |

#### PrEP Education (Psychoeducation) & TEAMS

#### Forms of PrEP & PrEP Safety

Did you know there are different forms of PrEP? PrEP can be a **pill** you take every day or by getting an **injection** every two months.

Also, the medications used for PrEP are used for to treat individuals living with HIV. Many patients report being anxious about taking PrEP due to long term side effects, however, **since** 

these medications have been used for years to treat HIV, we know the long term side effects, if any, are mild. In PrEP clinical trials, most people had no serious side effects. However, some people experienced mild side effects such as:

- upset stomach
- headache
- vomiting
- loss of appetite
- a small weight gain
- a change in the amount of some types of fats (lipids) in their blood

These side effects usually fade during the first month of taking PrEP.

How did learning about or hearing the side effects of PrEP make you feel? (scared? nervous? excited?)

Did hearing the side effects make you think about PrEP any differently? If so, how?

Sometimes people get nervous when considering a new medication.

Regardless of how you felt, all experiences are normal when considering taking a new medication. The key is to remember that if you believe taking PrEP may be in line with your values, these experiences are part of the process of living your best life.

Another way to think about this, is thinking back to when you asked your partner out for the very first time. How did you feel? Usually, people feel anxious when approaching partners for the first time. This is very normal and in the end is worth forming a meaningful connection.

The main takeaway messages from this section are that:

- There are different forms of PrEP, pill and injection.
- PrEP medications are not new, so we know most of the longer-term side effects.
- Most side effects of PrEP go away.
- Sometimes we experience unwanted emotions such as anxiety when doing new things that are important to us.

Now we are going to do an exercise to learn more about controlling emotions.

#### Lack of Control: Emotion Machine (Acceptance)

I want you to imagine that you are in this office with me. Imagine I have seated you in a big red chair and hooked you up to a giant metal machine. The machine has lots of buttons and wires. I strap your arms and legs to the machine and connect these wires to your head and chest. You are all plugged in. This machine can tell me exactly what you are thinking and feeling. Now I want you to think of anything but a red elephant. Okay? If you think of a red elephant, I am going to hit you with this book. So, think of anything but that. What are you thinking of? (usually a red elephant OR the thought of trying not to think of a red elephant) Okay, so we have now learned you are not always in control of what you think. Now I am going to ask you to not feel anxious.

You can feel anything other than anxiety... happiness, sadness, anger... just don't feel anxious. If you do, I am going to shoot you in the foot with this gun. What are you experiencing right now? (usually anxiety) Now we have learned that you are also not in control of emotions or thoughts.

Knowing this is helpful when trying to do things that are important to you but that make you feel or think in a way you don't want. Often times we try to control our emotions and thoughts and it ends up making them worse. However, if we notice these experiences without trying to change them, they can be more manageable.

# Cost of Avoiding Emotions Related to PrEP: Select Between 2 Lives (Acceptance) Long time vs. short time

In life there are two different kinds of lives to live.

In one life people are free from discomfort and anxiety. However, in this life people also do not have joy, happiness, or meaning in their life. People who pick this life usually do things to keep from feeling anything at all. Like using drugs excessively.

The second life people have discomfort and anxiety but also have joy, happiness, and meaning in their life. They do things that are important to them even though it may cause stress or discomfort.

Which life would you pick?

Truly living means that you experience the full range of emotions.

Another thing to think about is that many people avoid short term discomfort which often leads to long term discomfort. For example, someone may be aware that they need to get a flu shot but avoid it because they are afraid of shots. In the moment, they were able to avoid feeling the discomfort of getting a shot but put themselves at risk for getting the flu.

It is normal to not want to experience discomfort but sometimes this can have great costs like getting the flu, diabetes, or even HIV. PrEP is similar. Many people who know they may be at risk for HIV, do not want to experience the discomfort, shame, anxiety, fear, worry, or other types of emotional pain of going to a clinic appointment or taking a daily medication. However, avoiding these short term discomforts could have lifelong consequences.

Sometimes being willing to experience discomfort in the short term can save one from having to experience a lot more discomfort in the long-term.

#### Put up two fists to indicate each life.

Does this make sense to you? If you had to choose just one of these lives to live which life, would you choose?

Allow Patient to Respond.

Noticing discomfort and anxiety as part human experiences instead of trying to avoid them, actually helps you live more intentional and a fuller life.

For example, often times people with social anxiety will report that they don't want to go to a party. But if we peel this situation back like an onion and look under the surface we usually find that the person actually does want to attend the party and connect with others but do not want to experience the anxiety leading up to getting to the party.

The main takeaway messages from this section are that:

- Trying to avoid our emotions is not helpful.
- Sometimes being willing to experience discomfort in the short term can save one from having to experience a lot of discomfort in the long-term.

#### Singing Thoughts: Coping with Anxious Thoughts (Defusion)

- Let's talk about a fun way to cope with anxious thoughts. When was the last time you were anxious? Can you think of a specific thought you were having? (provide examples if needed: "everything is going to go bad" "what if people don't like me") Do you remember how anxious the thought made you at the time from 0-10, with 10 being super anxious?
- Okay, now I want you to do something super silly with me. We are going to sing that thought. (offer to sing with patient if they are unwilling, or sing for them if they are really resistant)(sing the thought a few times).
- Now that we have made a song out of that thought how anxious does the thought make you from 0-10?
- Usually, anxiety decreases when we spent some time noticing the thought is not something to be scared of. It won't jump out and get you (humor). Feel free to use this in the future to help with anxious thoughts if you found it helpful.

#### Coping with Emotions Using Senses (Present Moment Awareness)

One way to cope with emotions instead of avoiding them is to practice being in the moment. Let me know you an example of what this looks like.

Start by taking a few deep breaths. Inhale and exhale.

Next, I would like you to name all the colors you can find in this room. [allow time for response]

Now name one thing you can taste. This may be something you ate or drank recently. [allow time for response]

Now I would like you to check in with yourself and describe how you are feeling. Are you tired, awake, sad, happy, cold, hot? You could be feeling many different things. Take a minute to describe how all the things you are feeling. [allow time for response]

Now just take 3 more deep breaths. Notice how describing these things can be helpful to bring you back to the moment.

| T 1 | | ~~ | • |
|-----|------------|----|-------|
| HMA | $\alpha$ 1 | | CCIAN |
| Lnu | (// | DE | ssion |
| | , | | ~~~~ |

| Thank you for engaging in today's session. I would like you to review the values you identified once a week until we meet again. [Provide participant with their list of values and action items.] Your next appointment will be |
|---|
| Note: Please record action items for each participant. We will use them in next session. |
| Session Three |
| Session 3 Outline (45 minutes) 1Review previous session [5 minutes] 2.Dimensions of Sexuality (Psychoeducation, Acceptance) [10 minutes] 3.Influential People and Aspired Qualities (Values) [5 minutes] 4.Health of Others-Putting on Your Mask First (Values) [5 minutes] 5.Annoying Friend at Party: Alternative to Controlling Thoughts and Emotions [5 minutes] 6.Car Self-Worth Metaphor (Acceptance, Compassion, Self as Context) [5 minutes] 7.Honoring Past, Present, and Future Peers Exercise (Values and Perspective Taking) [5 minutes] 8.Summarize Session & Feedback [5 minutes] |
| Review Previous Session |
| Welcome back! To get started, I just want to briefly review a few things from previous sessions. You identified (say their values) as your values. Does that still seem accurate now that you have had time to think about things? Is there anything you would change? |
| You selected 3 action plan items to do that are in line with your values. How did that go? [Help participant problem solve if they were unable to complete the action plan] |
| How did that may you feel to complete (or not complete) the[action plan items]? |
| Action Plan |
| Similar to our last session, can you think of 3 action steps you can take that are in line with your values (list their values here)? These can be similar to the plans you listed in the last session or new ones. |
| 1 |

2.\_\_\_\_\_

3.\_

# Dimensions of Sexuality: Education on How Sexuality Develops (Psychoeducation & Acceptance)

We want to briefly discuss sexuality and how it is developed. Lots of people are uncomfortable talking about sex and when their mind creates graphic sexual images they try to control, avoid, or eliminate those pictures. But sex is actually a good thing, and we want to help you feel more comfortable talking about sex and to understand how sexuality is developed. All humans are sexual beings from birth.

Sex comes from the term "sexuality" that refers to all dimensions of being a sexual creature. These dimensions INFLUENCE and do not DETERMINE SEXUAL IDENTITY. As long as individuals are consenting adults, there are no good nor bad sexual preferences.

#### Briefly discuss each dimension.

- ⇒ **Biological:** Genetics, the body parts each of us have, and hormones all play a role in someone's sexuality.
  - For example, having a vagina and the worry about pregnancy, will cause you to have a different mental framework compared to someone who doesn't.
- ⇒ **Social:** Family impact and role models for all things sexual.
  - Think of your own parents, do you have a mom and dad, two moms, two dads, one parent only? Other family members also have an impact. You learn to be a sexual man, women, or couple from observing your family over time in thousands of sexual satiations that may not seem like they are sexual. For example, the way your family prepared and cleaned up after dinner may have an impact.
- ⇒ Cultural: Beliefs, values, behavior patterns, race, ethnicity, socioeconomic status, and physical environment.
  - For example, race and ethnic heritage transmit sexual information passed down through traditions that extend back hundreds of years. This also includes your coworkers, casual friends, and sexual partners all influence your sexuality.
  - For example, men have been known as the Breadwinners, while women have been the child caretakers.

#### ⇒ Political, Legal, Economic:

- Think of your sexuality like a board game. You and all the people in your life are the players and pieces. The board and the rules are the legal/political/economical dimensions.
- Examples of this include sex education in schools, laws regarding abortion, and prostitution can all have an impact.

#### ⇒ Psychological:

• *Thoughts and feelings all shape your sexuality over time.* 

In summary, sexuality is developed via nature and nurture. Some of your sexual preferences are influenced by biological things like genes, while others are influenced directly by your environment. The reason this study is targeting young Black men who have sex with men is because the rates of HIV are higher among this population, particularly in Mississippi. This is no one's fault, some people are just at higher risk due to sexual preferences and geographic location. It is important to note that humans do not pick their sexual identity and actually have little control over what their sexual preferences are.

Does all of this make sense? Do you have any questions?

#### **Influential People and Aspired Qualities (Values)**

Think about your heroes or people you look up to. Consider people who have inspired you: family members, friends, coaches, authors, artists, celebrities, or even fictional characters. PICK ONE Who would you most like to be like? Who is this person? [allow time for response] Now think about all the qualities you really admire in this person—not the person's circumstances, but personal qualities (i.e., kindness, strength) [allow time for discussion, take note of qualities].

How might these qualities translate into SOMEONE'S decision to take PrEP? [allow time for discussion]

#### Health of Others – Putting on Your Mask (Values)

Have you ever ridden in a plane before? What do they tell you when describing what to do if you need to put a mask on? Why do they tell you to put your mask on first? Right, in order to keep others safe sometimes we need to put our own mask on first.

How might taking PrEP be like putting on your mask in a plane? [allow time for discussion about how PrEP is a way to protect others in the community.]

Taking PrEP is like putting on your mask on a plane. You are first taking care of yourself and getting the protection you need and THEN you are offering to help protect others. Does this make sense? (answer any questions they may have)

#### Annoying Cousin at Party: Alternative to Controlling Thoughts and Emotions (Acceptance)

"Our next exercise is going to focus on how to handle thoughts and emotions. I want you to imagine you are throwing a huge party to celebrate your birthday at your house. What would the party theme be, what would be decorations be like, what would you wear? [allow time for response] Now I want you to imagine that you are at this party having a great time with your friends. Soon after the party starts your annoying cousin (who your mom forced you to invite) shows up at the party. They come into the party and start being loud and annoying so you decide to try to get them to leave. You finally get them to leave but a few minutes later they come back. Again, you work to get them to leave but they just keep coming back. Before you know it, the party is over, and people are leaving. You realize you spent most of the party trying to get your cousin to leave. What might your experience at the party be like if you had just decided to let your cousin stay? (would you have been able to enjoy some of the party even while they were being annoying)

Trying to control our emotions and thoughts looks similarly. Often, we are trying so hard to control these experiences that we are unable to enjoy life or engage in values driven behaviors. The alternative is to be honest with ourselves and make room for what we think and feel, even if these experiences are unpleasant.

Another way to think of this, imagine someone accidently drops half of your birthday cake on the ground. You can decide to be angry that you are missing half the birthday cake or acknowledge your sadness at missing half the birthday cake while also enjoying the other half of the cake.

#### Car Self-Worth Metaphor (Acceptance, Compassion, and Self as Context)

In this next exercise we are going to talk about how to view your body in a different way. Often people think that their body is what makes up who they are instead of the vessel used to carry ourselves. Another way to consider this is to image your body is a car and you are the person driving the car. Two separate things. You can turn the wheel of the car to change directions and feel the comfort of the seat, but you are not the car. You can also give the car an oil change and paint job to take care of it, but the person sitting inside the car stays the same. The worth of the person sitting inside the car is not dependent on how our "car" looks or functions. Similarly, how attractive or healthy we are does not impact our worth. The person inside your body is always worthy of love and kindness.

#### Honoring Past, Future, and Present Peers Exercise (Values and Perspective Taking)

We are going to do a brief exercise now. I am going to ask you a series of questions, but you don't need to answer them out loud. We will discuss at the end.

Take a few deep breaths. Slowly close your eyes.

#### Past

Imagine you are alive in the time before medications to treat HIV are available. Imagine many of your friends, peers, and past partners have been diagnosed with HIV, except there are no medications available to treat HIV yet. Imagine what emotions you might be experiencing if this happened? (PAUSE)

#### **Future**

Now I want you to imagine you are alive 100 years from now in the future. Image what it would be like if HIV no longer existed. Imagine what this would feel like. (PAUSE) What do you think you would say to people who had taken PrEP or their HIV medications to eliminate HIV in the world? Do you think you would thank them? What exactly do you think you would say? [PAUSE]

Take another deep breath.

#### Now

Now imagine you back to present day. What might you say to your peers living with HIV about taking their medication. What might you say to your peers at risk for HIV about PrEP? [PAUSE] Would you encourage them to their medication or to take PrEP? Would you warn them about how serious HIV can be when untreated? Would you inform them about how PrEP can prevention HIV?

Take a few more deep breaths. When you are ready you may open your eyes.

How was that? What did you feel?

Some patients have reported that taking PrEP allows them to honor those who have passed or who have been impacted by HIV. Does this resonate with you? [allow time to respond]

# End of Session

Over the past three sessions we have talked a lot about PrEP, values, and how to cope with unhelpful thoughts and feelings. How motivated are you to take PrEP after these discussions? Have these conversations been helpful in linking your values to taking PrEP? How so? Is there anything you would change about any of the sessions?

Thank you for your feedback and for participating in this study.

Note: Please record intervention feedback from the participants.

# Values Inventory and Action Plan Sheet

| | Identified Values |
|----|-------------------|
| 1 | |
| 1 | |
| 2 | _ |
| 3 | _ |
| 4 | |
| 5 | - |
| | Action Plan |
| 1. | |
| 2 | |
| 2 | |

| ACTPrEP Session One Checklist | | | |
|---|---|---|---|
| Content | Completed | Not<br>Completed | Reason Not<br>Completed |
| Primary Values Exercise | | | |
| PrEP Education | | | |
| Compared PrEP to Other Medications | | | |
| Carrying Weight Metaphor: Control in Reducing HIV Risk | | | |
| Discuss Barriers to PrEP Use: Finding a PrEP Provider | | | |
| Discuss Barriers to PrEP Use: Transportation | | | |
| Discuss Barriers to PrEP Use: Paying for PrEP Appointments | | | |
| Discuss Barriers to PrEP Use: Paying for PrEP Medication | | | |
| Coffee Cup Experiential Exercise | | | |
| 5-Year-Old Self Exercise | | | |
| Created an Action Plan | | | |
| Wrote Participants Values Down | | | |
| Scheduled Next Session | | | |

| ACTPrEP Session Two Checklist | | | |
|---|---|---|---|
| Content | Completed | Not<br>Completed | Reason Not<br>Completed |
| Reviewed Previous Session | | | |
| Created an Action Plan | | | |
| PrEP Education & TEAMS Discussion | | | |
| Discussed Different Forms of PrEP | | | |
| Discussed PrEP Safety and Explained Use for HIV | | | |
| Lack of Control: Emotion Machine Exercise | | | |
| Cost of Avoiding Emotions Related to PrEP: 2 Lives | | | |
| Singing Thoughts Exercise | | | |
| Coping with Emotions Using Senses Exercise | | | |
| Wrote Participants Values Down | | | |
| Scheduled Next Session | | | |

| ACTPrEP Session Three Checklist | | | |
|---|---|---|---|
| Content | Completed | Not<br>Completed | Reason Not |
| Reviewed Previous Session | | | |
| Create Action Plan | | | |
| Dimensions of Sexuality | | | |
| Influential People and Aspired Qualities | | | |
| Health of Others-Putting on Your Mask First | | | |
| Cousin at Party: Alternative to Controlling | | | |
| Car Self-Worth Metaphor | | | |
| Honoring Past, Present, and Future Peers Exercise | | | |
| Feedback on Intervention | | | |

### **Enhanced Standard of Care (ESOC) Intervention**

| Session Content |
|--------------------------------------------------------|
| Session 1 Outline (60 minutes) |
| 1.Introduce self, review goal of study, review |
| confidentiality [5 minutes] |
| 2.Self-Care Discussion [5 minutes] |
| 3.PrEP Education (Psychoeducation) [5 minutes] |
| 4.HIV and PrEP Rates (Psychoeducation) [5 minutes] |
| 5.Discuss Structural Barriers to PrEP Use [10 minutes] |
| 6.Summarize session [5 minutes] |
| Session 2 Outline (30 minutes) |
| 1.Self-Care Discussion (5 minutes) |

- 2. Review Previous Session Content (5 minutes)
- 3. Considered PrEP Discussion (5 minutes)
- 4. Review Barriers (5 minutes)
- 5.End of Session (5 minutes)

# Session 3 Outline (30 minutes)

- 1.Self-Care Discussion (5 minutes)
- 2. Review Previous Session Content (5 minutes)
- 3. Considered PrEP Discussion (5 minutes)
- 4. Review Barriers (5 minutes)
- 5.End of Session (5 minutes)

| Session<br>Number | Key Message |
|---|---|
| Session<br>One | <ul> <li>Provide Brief PrEP Psychoeducation</li> <li>Identify &amp; Address Barriers to PrEP<br/>Use</li> </ul> |
| Session<br>Two | <ul><li>Review PrEP Psychoeducation</li><li>Review Barriers to PrEP</li></ul> |
| Session<br>Three | <ul><li>Review PrEP Psychoeducation</li><li>Review Barriers to PrEP</li></ul> |

#### **Intervention Manual**

#### **Session One**

#### **Session 1 Outline (60 minutes)**

- 1. Introduce self, review goal of study, review confidentiality [10 mins]
- 2.Self-Care Discussion [5 minutes]
- 3.PrEP Education [5 mins]
- 4.HIV and PrEP Rates [5 minutes]
- 5. Discuss Barriers to PrEP Use [10 minutes]
- 6.Summarize session [5 minutes]

#### **Introductions**

- Introduce yourself and your job/role.
- Share some information about how this work is meaningful to the interventionist, perhaps a piece of personal history regarding this work or the value of this work to the interventionist.
- Thank the participant for participating in the study.
- Review the goal of the study.
- Remind participant that of confidentiality and its limits.

Hi, my name is \_\_\_\_ and I work as a \_\_\_ at \_\_\_ . Thank you for completing the survey and for your willingness to participate in this study session. The goal of this study is to help you understand PrEP more and to help eliminate any barriers to PrEP use. Anything you say during this meeting will be kept confidential and not shared with anyone else. The only exception to this is if you report thoughts with an intent and plan of harming yourself or someone else. If you report those things, I will need to notify others so that we can keep everyone safe.

We will be audio recording these sessions so that our study team can be sure I covered all the topics. All recordings are saved on a secure drive and will not be linked back to your name. Once they have checked the recordings they will be deleted. Any questions before we get started?

#### Self-Care Discussion

#### **What is Self-Care**

Do you know what self-care is? [allow time for participant to respond]

Self-care is when individuals look after their own health using the knowledge and resources available to them. There are five different types of self-care: physical, emotional, psychological, spiritual and professional care.

#### **Self-Care Strategies**

Do you do anything for self-care? [allow time for participant to respond]

There are lots of ways people engage in self-care. There are no right or wrong ways as long as you are caring for yourself. Self-care can include making healthy food choices, exercising, getting plenty of sleep, and going to healthcare providers like your dentist or primary care doctor for checkups.

#### PrEP Education (Psychoeducation)

#### **Assess Participant Experience with PrEP**

Do you know what PrEP is or have you ever considered taking PrEP? [allow time for participant to respond]

#### **What is PrEP**

PrEP stands for preexposure prophylaxis. PrEP prevents HIV infection from spreading if you are exposed to the virus. This is done by either taking a pill every day or by getting an injection every two months. There are currently three drugs used for PrEP. Truvada, Descovy, and Cabotegravir are medications used to treat individuals living with HIV, and ALSO used as forms of PrEP to prevent HIV from spreading to someone who is HIV negative. Truvada or Descovy are the oral/pill form of PrEP and Cabotegravir is the injectable form of PrEP. Descovy and Cabotegravir are not prescribed for women (persons assigned female at birth).

If you were to take PrEP, would you take a pill or the injectable? Why?

#### Is PrEP Safe

These are the same medicines that are highly effective at stopping the virus from growing in those living with HIV. In fact, individuals living with HIV who take these medications as prescribed can have undetectable amounts of HIV in their blood and are unable to transmit HIV to others. This is known as U=U or U ndetectable = U ntransmittable. Since these medications have been used for years to treat HIV, we know the long-term side effects are mild. In P reclinical trials, most people had no serious side effects. However, some people taking oral P resperienced early side effects such as:

- upset stomach
- headache
- vomiting
- loss of appetite
- a small weight gain
- a change in the amount of some types of fats (lipids) in their blood

These side effects usually fade during the first month of taking PrEP.

Many people in trials of PrEP injections had a reaction at the injection site like mild pain, redness, or swelling. These reactions were mild and lasted only a couple of days.

#### Why Take PrEP

Nearly 40,000 people get infected with HIV each year in the U.S. More of these infections are happening in some groups of people and some areas of the country than in others. Mississippi is among the states with the highest rates of new HIV infections. You should consider taking PrEP if: You sometimes have sex without using a condom OR

- You have recently been told by a health care provider that you had a sexually transmitted infection OR
- If your partner has HIV infection OR
- If you are sexually active in an area with higher rates of HIV infection OR
- *Use injection drugs recreationally*

#### Who Should Take PrEP

Anyone at risk for HIV can benefit from PrEP.

#### HIV and PrEP Rates (Psychoeducation)

Now we are going to briefly discuss the rates of PrEP use among people in the United States.

- The number of PrEP users in the U.S. increased by 23% from 2020 to 2021.
- However, the South accounted for 52% of HIV diagnoses but only accounted for 39% of PrEP users.
- Among all PrEP users in the U.S., 92% were male and only 8% were female, even though women comprised 18% of new HIV diagnoses.
- Black people represented 14% of PrEP users, but 42% of new HIV diagnoses.
- Regionally, Black individuals made up 52% of new HIV diagnoses in the South, but only 21% of PrEP users in the South.
- Of the 7 states with the greatest unmet need for PrEP among Black people, three were in the South: Arkansas, Mississippi, and Alabama.
- There is a high need for more individuals to take PrEP, Especially, women, Black individuals, and individuals living in Mississippi.

#### Barriers to PrEP Use

Can you think of anything that would get in the way of you being able to take PrEP if you decided to get a prescription? (allow patient to respond first and then explore each barrier below) [document which barriers the participant anticipates]

| Barrier | PrEP Resources |
|---|---|
| Finding a Doctor to<br>Prescribe PrEP | d. Open Arms Healthcare Center<br>805 E River Pl Jackson, Mississippi 39202<br>(601) 500-7660 |
| | e. Express Personal Health Jackson Medical Mall, 350 W. Woodrow Wilson Avenue. Third Floor 601-815-5861; eph@umc.edu |
| | f. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP) |
| | Primary Care Providers. |
| | i. Dr Arenia C Mallory Community Health Center |
| | 276 Nissan Pkwy Canton, Mississippi 39046<br>(601) 859-1798 |
| | j. GA Carmichael Family Health Center |
| | 1547 Jerry Clower Blvd Yazoo City, Mississippi 39194<br>(662) 746-6532 |
| | k. GA Carmichael Family Health Center |
| | 1668 W Peace St Canton, Mississippi 39046 |

| | (601) 859-5213 |
|---|---|
| | l. Jackson-Hinds Comprehensive Health Center<br>514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216 |
| | (601) 362-5321<br>m. AIDS Healthcare Foundation |
| | 766 Lakeland Dr Jackson, Mississippi 39216 (601) 368-3440 |
| | n. TIN Rx 2657 Lakeland Dr Jackson, Mississippi 39232 (601) 588-2490 |
| | o. Quinn Healthcare PLLC 768 Avery N Blvd Ridgeland, Mississippi 39157 (601) 487-6482 |
| | p. Southern Medical Care 6600 US Highway 98, Hattiesburg, MS 39402 (601)-261-2727 |
| | Local Health Department (can do labs and set you up with Telehealth appointment for PrEP) |
| | You can search for providers on this website: <a href="https://www.pleaseprepme.org">https://www.pleaseprepme.org</a> |
| Telehealth Services | a. Jackson-Hinds Comprehensive Health Center<br>514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216<br>(601) 362-5321 |
| | b. Dr Arenia C Mallory Community Health Center<br>276 Nissan Pkwy Canton, Mississippi 39046<br>(601) 859-1798 |
| | c. Open Arms Healthcare Center<br>805 E River Pl Jackson, Mississippi 39202<br>(601) 500-7660 |
| | d. Dr Arenia C Mallory Community Health Center |
| | 276 Nissan Pkwy Canton, Mississippi 39046<br>(601) 859-1798 |
| | e. Southern Medical Care<br>6600 US Highway 98, Hattiesburg, MS 39402<br>(601)-261-2727 |
| Transportation to<br>Clinic Appointments | <ul> <li>a. Open Arms can provide transportation to appointments as long as you call and pre-schedule with the clinic.</li> <li>b. Express Personal Health does not offer transportation.</li> </ul> |
| Paying for PrEP | Express Personal Health visits and labs are free. |

| | Local Health Department (can do labs and set you up with Telehealth appointment for PrEP- Free Services) |
|---|---|
| Paying for PrEP<br>Medication | a. Mississippi Family Planning Waiver can cover the cost of PrEP. b. Gilead Payment Assistant Program can also help cover the cost of PrEP: https://www.am10.gilead.com/en/purpose/medication-access |
| PrEP Mailing Services | a. Jackson-Hinds Comprehensive Health Center<br>b. GA Carmichael Family Health Center<br>c. Open Arms Healthcare Center<br>d. Dr. Arenia C. Mallory Community Health Center<br>e. CVS<br>f. Walgreens |

#### End of Session

Thank you for engaging in today's session. Do you have any questions about anything that we covered today?

Your next appointment will be . .

Note: Please record barriers for each participant.

#### **Session Two**

#### Session 2 Outline (30 minutes)

- 1.Self-Care Discussion (5 minutes)
- 2. Review Previous Session Content (5 minutes)
- 3. Considered PrEP Discussion (5 minutes)
- 4. Review Barriers (5 minutes)
- 5.End of Session (5 minutes)

#### Self-Care Discussion

#### **Self-Care Strategies**

Before we talk about PrEP, I just want to check in to see if you were able to do anything for self-care in the past week? [allow time for participant to respond]

Remember, there are lots of ways people engage in self-care. Self-care can include making healthy food choices, exercising, getting plenty of sleep, and going to healthcare providers like your dentist or primary care doctor for checkups.

#### **Review Previous Session Content**

Can you tell me what you remember from our last discussion?

Great, now I am going to briefly review what we discussed in our last meeting.

# **Review Each of the Concepts Below What is PrEP**

PrEP stands for preexposure prophylaxis. PrEP prevents HIV infection from spreading if you are exposed to the virus. There are currently three drugs used for PrEP. Truvada, Descovy, and Cabotegravir. Truvada or Descovy are the oral/pill form of PrEP and Cabotegravir is the injectable form of PrEP. Descovy and Cabotegravir are not prescribed for women (persons assigned female at birth).

#### Is PrEP Safe

In PrEP clinical trials, most people had no serious side effects. However, some people taking oral PrEP experienced early side effects such as:

- upset stomach
- headache
- vomiting
- loss of appetite
- a small weight gain
- a change in the amount of some types of fats (lipids) in their blood

These side effects usually fade during the first month of taking PrEP.

### Why Take PrEP

Nearly 40,000 people get infected with HIV each year in the U.S. More of these infections are happening in some groups of people and some areas of the country than in others. Mississippi is among the states with the highest rates of new HIV infections. You should consider taking PrEP if:

- You sometimes have sex without using a condom OR
- You have recently been told by a health care provider that you had a sexually transmitted infection OR
- If your partner has HIV infection OR
- If you are sexually active in an area with higher rates of HIV infection OR
- *Use injection drugs recreationally*

#### Who Should Take PrEP

Anyone at risk for HIV can benefit from PrEP.

#### HIV and PrEP Rates (Psychoeducation)

- The number of PrEP users in the U.S. increased by 23% from 2020 to 2021.
- However, the South accounted for 52% of HIV diagnoses but only accounted for 39% of PrEP users.
- Among all PrEP users in the U.S., 92% were male and only 8% were female, even though women comprised 18% of new HIV diagnoses.
- Black people represented 14% of PrEP users, but 42% of new HIV diagnoses.
- Regionally, Black individuals made up 52% of new HIV diagnoses in the South, but only 21% of PrEP users in the South.
- There is a high need for more individuals to take PrEP. Especially, individuals living in Mississippi.

#### **Considered PrEP Discussion**

- Have you thought about getting a prescription for PrEP since our last meeting?
- Do you think PrEP could be a useful medication for you? Why or why not.

### **Review Barriers**

If you were to decide to get a prescription for PrEP, do you anticipate there being any barriers to you being able to get a prescription?

| Barrier | PrEP Resources |
|---|---|
| | g. Open Arms Healthcare Center |
| Finding a Doctor to<br>Prescribe PrEP | 805 E River Pl Jackson, Mississippi 39202 |
| rescribe 1 TE1 | (601) 500-7660<br>h. Express Personal Health |
| | Jackson Medical Mall, 350 W. Woodrow Wilson Avenue. |
| | Third Floor |
| | 601-815-5861; <u>eph@umc.edu</u> |
| | i. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP) |
| | Primary Care Providers. |
| | q. Dr Arenia C Mallory Community Health Center |
| | 276 Nissan Pkwy Canton, Mississippi 39046 |
| | (601) 859-1798 |
| | r. GA Carmichael Family Health Center |
| | 1547 Jerry Clower Blvd Yazoo City, Mississippi 39194<br>(662) 746-6532 |
| | s. GA Carmichael Family Health Center |
| | 1668 W Peace St Canton, Mississippi 39046<br>(601) 859-5213 |
| | t. Jackson-Hinds Comprehensive Health Center |
| | 514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216<br>(601) 362-5321 |
| | u. AIDS Healthcare Foundation |
| | 766 Lakeland Dr Jackson, Mississippi 39216<br>(601) 368-3440 |
| | v. TIN Rx |
| | 2657 Lakeland Dr Jackson, Mississippi 39232<br>(601) 588-2490 |
| | w. Quinn Healthcare PLLC |
| | 768 Avery N Blvd Ridgeland, Mississippi 39157<br>(601) 487-6482 |
| | x. Southern Medical Care |
| | 6600 US Highway 98, Hattiesburg, MS 39402<br>(601)-261-2727 |
| | Local Health Department (can do labs and set you up with Telehealth appointment for PrEP) |

| | You can search for providers on this website: <a href="https://www.pleaseprepme.org">https://www.pleaseprepme.org</a> |
|---|---|
| Telehealth Services | a. Jackson-Hinds Comprehensive Health Center 514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216 (601) 362-5321 b. Dr Arenia C Mallory Community Health Center 276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798 c. Open Arms Healthcare Center 805 E River Pl Jackson, Mississippi 39202 (601) 500-7660 d. Dr Arenia C Mallory Community Health Center 276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798 e. Southern Medical Care 6600 US Highway 98, Hattiesburg, MS 39402 (601)-261-2727 |
| Transportation to<br>Clinic Appointments | <ul> <li>a. Open Arms can provide transportation to appointments as long as you call and pre-schedule with the clinic.</li> <li>b. Express Personal Health does not offer transportation.</li> </ul> |
| Paying for PrEP<br>Appointments | Express Personal Health visits and labs are free. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP- Free Services) |
| Paying for PrEP<br>Medication | a. Mississippi Family Planning Waiver can cover the cost of PrEP. b. Gilead Payment Assistant Program can also help cover the cost of PrEP: https://www.am10.gilead.com/en/purpose/medication-access |
| PrEP Mailing Services | a. Jackson-Hinds Comprehensive Health Center<br>b. GA Carmichael Family Health Center<br>c. Open Arms Healthcare Center<br>d. Dr. Arenia C. Mallory Community Health Center<br>e. CVS<br>f. Walgreens |

End of Session

Thank you for engaging in today's session. Do you have any questions about anything that we covered today?

| Your next appointment will be |
|-------------------------------|
|-------------------------------|

Note: Please record barriers for each participant.

#### **Session Three**

#### Session 3 Outline (30 minutes)

- 1.Self-Care Discussion (5 minutes)
- 2. Review Previous Session Content (5 minutes)
- 3. Considered PrEP Discussion (5 minutes)
- 4. Review Barriers (5 minutes)
- 5.End of Session (5 minutes)

#### Self-Care Discussion

#### **Self-Care Strategies**

Before we talk about PrEP, I just want to check in to see if you were able to do anything for self-care in the past week? [allow time for participant to respond]

Remember, there are lots of ways people engage in self-care. Self-care can include making healthy food choices, exercising, getting plenty of sleep, and going to healthcare providers like your dentist or primary care doctor for checkups.

#### **Review Previous Session Content**

Can you tell me what you remember from our last discussion?

Great, now I am going to briefly review what we discussed in our last meeting.

# Review Each of the Concepts Below

#### What is PrEP

PrEP stands for preexposure prophylaxis. PrEP prevents HIV infection from spreading if you are exposed to the virus. There are currently three drugs used for PrEP. Truvada, Descovy, and Cabotegravir. Truvada or Descovy are the oral/pill form of PrEP and Cabotegravir is the injectable form of PrEP. Descovy and Cabotegravir are not prescribed for women (persons assigned female at birth).

#### Is PrEP Safe

In PrEP clinical trials, most people had no serious side effects. However, some people taking oral PrEP experienced early side effects such as:

- upset stomach
- headache
- vomiting
- loss of appetite
- a small weight gain
- a change in the amount of some types of fats (lipids) in their blood

These side effects usually fade during the first month of taking PrEP.

#### Why Take PrEP

Nearly 40,000 people get infected with HIV each year in the U.S. More of these infections are happening in some groups of people and some areas of the country than in others. Mississippi is among the states with the highest rates of new HIV infections. You should consider taking PrEP if:

- You sometimes have sex without using a condom OR
- You have recently been told by a health care provider that you had a sexually transmitted infection OR
- If your partner has HIV infection OR
- If you are sexually active in an area with higher rates of HIV infection OR
- If you use injection drugs recreationally

#### Who Should Take PrEP

Anyone at risk for HIV can benefit from PrEP.

#### HIV and PrEP Rates (Psychoeducation)

- The number of PrEP users in the U.S. increased by 23% from 2020 to 2021.
- However, the South accounted for 52% of HIV diagnoses but only accounted for 39% of PrEP users.
- Among all PrEP users in the U.S., 92% were male and only 8% were female, even though women comprised 18% of new HIV diagnoses.
- Black people represented 14% of PrEP users, but 42% of new HIV diagnoses.
- Regionally, Black individuals made up 52% of new HIV diagnoses in the South, but only 21% of PrEP users in the South.
- There is a high need for more individuals to take PrEP. Especially, individuals living in Mississippi.

#### **Considered PrEP Discussion**

- Have you thought any about getting a prescription for PrEP since our last meeting?
- Do you think PrEP could be a useful medication for you? Why or why not.

#### **Review Barriers**

If you were to decide to get a prescription for PrEP, do you anticipate there being any barriers to you being able to get a prescription?

| Barrier | PrEP Resources |
|---|---|
| Finding a Doctor to<br>Prescribe PrEP | j. Open Arms Healthcare Center<br>805 E River Pl Jackson, Mississippi 39202<br>(601) 500-7660 |
| | k. Express Personal Health Jackson Medical Mall, 350 W. Woodrow Wilson Avenue. Third Floor 601-815-5861; eph@umc.edu |

l. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP)

#### Primary Care Providers.

y. Dr Arenia C Mallory Community Health Center

276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798

z. GA Carmichael Family Health Center

1547 Jerry Clower Blvd Yazoo City, Mississippi 39194 (662) 746-6532

aa. GA Carmichael Family Health Center

1668 W Peace St Canton, Mississippi 39046 (601) 859-5213

bb. Jackson-Hinds Comprehensive Health Center

514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216 (601) 362-5321

cc. AIDS Healthcare Foundation

766 Lakeland Dr Jackson, Mississippi 39216 (601) 368-3440

dd. TIN Rx

2657 Lakeland Dr Jackson, Mississippi 39232 (601) 588-2490

ee. Quinn Healthcare PLLC

768 Avery N Blvd Ridgeland, Mississippi 39157 (601) 487-6482

ff. Southern Medical Care

6600 US Highway 98, Hattiesburg, MS 39402 (601)-261-2727

Local Health Department (can do labs and set you up with Telehealth appointment for PrEP)

You can search for providers on this website: https://www.pleaseprepme.org

| Telehealth Services | a. Jackson-Hinds Comprehensive Health Center 514 A-B E Woodrow Wilson Dr Jackson, Mississippi 39216 (601) 362-5321 b. Dr Arenia C Mallory Community Health Center 276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798 c. Open Arms Healthcare Center 805 E River Pl Jackson, Mississippi 39202 (601) 500-7660 d. Dr Arenia C Mallory Community Health Center 276 Nissan Pkwy Canton, Mississippi 39046 (601) 859-1798 e. Southern Medical Care 6600 US Highway 98, Hattiesburg, MS 39402 (601)-261-2727 |
|---|---|
| Transportation to<br>Clinic Appointments | <ul> <li>a. Open Arms can provide transportation to appointments as long as you call and pre-schedule with the clinic.</li> <li>b. Express Personal Health does not offer transportation.</li> </ul> |
| Paying for PrEP<br>Appointments | Express Personal Health visits and labs are free. Local Health Department (can do labs and set you up with Telehealth appointment for PrEP- Free Services) |
| Paying for PrEP<br>Medication | a. Mississippi Family Planning Waiver can cover the cost of PrEP. b. Gilead Payment Assistant Program can also help cover the cost of PrEP: https://www.am10.gilead.com/en/purpose/medication-access |
| | a. Jackson-Hinds Comprehensive Health Center<br>b. GA Carmichael Family Health Center<br>c. Open Arms Healthcare Center<br>d. Dr. Arenia C. Mallory Community Health Center<br>e. CVS<br>f. Walgreens |

# End of Session

Thank you for engaging in today's session. Do you have any questions about anything that we covered today?

Thank you for participating to our study.

Note: Please record barriers for each participant.

| ESOC Session One Checklist | | | |
|---|---|---|---|
| Content | Completed | Not<br>Completed | Reason Not<br>Completed |
| Self-Care Discussion | | | |
| General PrEP Education | | | |
| HIV and PrEP Rates | | | |
| Discuss Barriers to PrEP Use: Finding a PrEP Provider | | | |
| Discuss Barriers to PrEP Use: Transportation | | | |
| Discuss Barriers to PrEP Use: Paying for PrEP Appointments | | | |
| Discuss Barriers to PrEP Use: Paying for PrEP Medication | | | |
| Scheduled Next Session | | | |

| ESOC Session Two Checklist | | | |
|---|---|---|---|
| Content | Completed | Not<br>Completed | Reason<br>Not<br>Completed |
| Self-Care Discussion | | | |
| Reviewed Previous Session | | | |
| Considered PrEP Discussion | | | |
| Review Barriers | | | |
| Scheduled Next Session | | | |

| ESOC Session Three Checklist | | | |
|---|---|---|---|
| Content | Completed | Not<br>Completed | Reason Not<br>Completed |
| Self-Care Discussion | | | |
| Reviewed Previous Session | | | |
| Considered PrEP Discussion | | | |
| Review Barriers | | | |
| Scheduled Next Session | | | |

#### **Analytic Plan**

Descriptive statistics (e.g., means, standard deviations, frequencies) will be calculated to summarize participant characteristics. Between-group differences (ACTPrEP vs ESOC Group) in baseline characteristics will be assessed using t-tests for continuous variables, chi-squared tests for categorical variables, and non-parametric tests as appropriate. Data will be aggregated across follow-up assessments (0, 6 weeks, 12 weeks) and analyzed using generalized linear models. We will test for differences in linear change over time between ACTPrEP and ESOC groups on each outcome variable. We will evaluate differences in the proportion of participants who engaged in PrEP (attended PrEP medical visit or fill a PrEP prescription at a pharmacy). We will obtain these data through patient chart review and pharmacy data. Propensity scores (i.e., inverse probability or treatment weighting) will be used to account for any imbalance in baseline characteristics between conditions.